CLINICAL TRIAL: NCT06121414
Title: Effectiveness of Combined Laserpuncture And Antiemetic Therapy on the Rhodes Index of Nausea, Vomiting and Reatching (RINVR) Scores in Adolescent Cancer Patients Undergoing Chemotherapy
Brief Title: Effectiveness of Laserpuncture and Standard Antiemetic on RINVR Scores in Adolescent Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ramadia Yunita, doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23061053
Record Dates: First submitted 2023-10-30; First posted 2023-11-08 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laserpuncture (Experimental): Laserpuncture using continous wave, 2 Joule in on condition
  Interventions: Device: laserpuncture
- Sham Laserpuncture (Sham Comparator): Sham laser using laserpuncture in off condition
  Interventions: Device: Sham Laserpuncture

INTERVENTIONS:
Device: laserpuncture — laserpuncture use continous wave,dose 2 Joule, 785nm, 50mw
  Arms: Laserpuncture
Device: Sham Laserpuncture — Sham laser using laserpuncture in off condition
  Arms: Sham Laserpuncture

SUMMARY:
Chemotherapy is a common treatment for treating cancer. Chemotherapy induced nausea and vomiting (CINV) is nausea and vomiting that occurs after chemotherapy. Complete protection of standard antiemetic drugs against CINV symptoms in children and adolescents receiving moderately and strongly emetogenic chemotherapy drugs was less than 50%.

The side effects of chemotherapy in the form of CINV are so unpleasant that chemotherapy causes extreme anxiety and stress. The psychological characteristics of adolescents who have a greater perception of the changes that occur cause more frequent anxiety which can increase the risk of CINV.

Acupuncture with laserpuncture modality is a non-pharmacological therapy that has a good effect on CINV symptoms in adolescents. This research was conducted for the first time in Brazil in 2019, while in Indonesia there has never been any research on this matter. So it is hoped that this research will be the first research in Indonesia to prove that the effect of laserpuncture plays a role in CINV symptoms in adolescents and can be an additional treatment in standard therapy for CINV problems in adolescents.

DETAILED DESCRIPTION:
This is a clinical trial study to evaluate and compare the effects of laserpuncture and sham laserpuncture as a therapy for Chemotherapy induced nausea and vomiting (CINV) . The subjects are 58 males/female and will be randomly assigned to 2 groups: (1) laserpunctur and (2) Sham laserpuncture. The outcome will be assessed before treatment (baseline), in chemotherapy procedure and 3 days after chemotherapy. Patients and the outcome assessors will be blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent cancer patients aged 10 - 18 years
2. Patients undergoing chemotherapy with moderate and/or strong emetogenic chemotherapy drugs
3. Patients with CINV and/or at risk of CINV
4. Willing to take part in research until completion
5. The patient has not received acupuncture therapy in the last 1 week

Exclusion Criteria:

1. Patients with cancerous lesions or ulcers at the location of the acupuncture points to be selected
2. Patients with digestive tract organ malignancies with complaints of nausea and vomiting before chemotherapy
3. Patients with unstable hemodynamic conditions

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Rhodes Index nausea, vomiting and Reatching Score (RINVR) | before chemotherapy, in chemotherapy procedure, 3 days after chemotherapy
  Score for measuring nausea, vomiting and reatching after chemotherapy. minimum score is 0 and maximum score is 32

OTHER OUTCOMES:
Screen for Child Anxiety Related Disorders (SCARED) | before Chemotherapy, 3 days after chemotherapy
  Score for measuring anxiety for Child. score 25 or more is anxiety. minimum score is 0 and maximum score is 82

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI KR RSCM, Principal Investigator — The Ethics Committee of the Faculty Of Medicine, University of Indonesia
Locations (2):
- Indonesia (2):
  - Dharmais Cancer, Hospital, Jakarta, DKI Jakarta
  - Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta

IPD SHARING:
Plan to Share IPD: No